CLINICAL TRIAL: NCT03967171
Title: The Comparison of the Effect of Different Oxytocin Administrations on the Blood Loss During Cesarean Delivery: a Randomised Controlled Trial
Brief Title: The Comparison of the Effect of Different Oxytocin Administrations on the Blood Loss During Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BezmialemVU Oxytocin effect
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Cesarean Section Complications; Postpartum Hemorrhage; Blood Loss, Surgical; Blood Loss, Postoperative; Postoperative Pain; Atony, Uterine
Keywords: Oxytocin; cesarean section; uterine atony; Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage; Blood Loss, Surgical; Postoperative Hemorrhage; Pain, Postoperative; Uterine Inertia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- before uterine incision oxytocin group (Experimental): IV infusion of 20 IU of oxytocin started before uterine incision
  Interventions: Other: before uterine incision oxytocin
- after clamping the umbilical cord oxytocin group (Active Comparator): IV infusion of 20 IU of oxytocin started immediately after clamping the umbilical cord
  Interventions: Other: after clamping the umbilical cord oxytocin

INTERVENTIONS:
Other: before uterine incision oxytocin — blood loss during elective cesarean section
  Arms: before uterine incision oxytocin group
Other: after clamping the umbilical cord oxytocin — blood loss during elective cesarean section
  Arms: after clamping the umbilical cord oxytocin group

SUMMARY:
This study compares the effect of starting intravenous oxytocin infusion early before uterine incision versus late after umbilical cord clamping on the blood loss during elective cesarean section

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is still the major cause of maternal morbidity and mortality worldwide contributing to nearly 25% of direct maternal deaths. The average blood loss during cesarean section is 1000 ml which is nearly double the blood loss during vaginal delivery. Worldwide, the most commonly used uterotonic for the prevention of PPH is oxytocin. Several regimens of oxytocin have been tested during cesarean section with variable wanted (uterotonic) and unwanted (cardiovascular) effects. In the current study, we tested the hypothesis that initiating IV oxytocin infusion earlier before uterine incision would induce a rapid acceptable uterine contraction and minimize the intraoperative blood loss than the same dose administered after delivery of the fetus.

ELIGIBILITY:
Inclusion Criteria:

* single fetus at term >37 weeks of gestational age

Exclusion Criteria:

* history of previous cesarean section
* history of previous uterine surgery
* multiple gestation, placenta previa, polyhydramnious, fetal macrosomia
* women at high risk for uterine atony such as anemia (Hb < 8 gm/dL)
* uterine atony history
* gestational diabetes mellitus, gestational hypertension, preeclampsia, current or previous history of heart disease, liver, renal disorders or known coagulopath

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 101 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
blood loss during elective cesarean section | 2 hours
  The intraoperative blood loss will be measured by adding the volume of the suction bottle with the blood soaked sponges (know dry weight). The blood loss was estimated after excluded amniotic fluid volume in the suction bottle in each case

SECONDARY OUTCOMES:
postoperative blood loss | 24 hours
  The hemoglobin and hematocrit values will be measured 24 hours after CS

OTHER OUTCOMES:
postoperative pain score | 24 hours
  The Visual Analogue Scale (VAS) will be implemented postoperative day 0 and postoperative 1st day
neonatal wellbeing | 2 hours
  Apgar scores (1 and 5 minutes) will be compared

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No